CLINICAL TRIAL: NCT04004689
Title: Use of the 6-minute Stepper Test to Individualise Pulmonary Rehabilitation in Patients With Severe to Very Severe Chronicle Obstructive Pulmonary Disease
Brief Title: 6-minute Stepper Test and Pulmonary Rehabilitation in Patients With Severe to Very Severe Chronicle Obstructive Pulmonary Disease
Acronym: 6STaR-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: 6STaR-2
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; 6-minute Stepper Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective observational cohort: Every patient referred to pulmonary rehabilitation program will be eligible. They will perform cardiopulmonary exercise testing prior to join the rehabilitation program.
  During the first session of pulmonary rehabilitation, they will perform 2 6-minute stepper test with a rest of 20 minutes minimum between each test.
  Interventions: Other: 2 times : 6-minute stepper test with a rest of 20min between each test.

INTERVENTIONS:
Other: 2 times : 6-minute stepper test with a rest of 20min between each test. — Patients will perform two 6-minute stepper tests separated by a rest period of at least 20 minutes. The second test will begin when the heart rate and the transcutaneous oxygen saturation values will be returned to baseline values. Standardization of the instructions for the test will be based on the actual guidelines for the 6-minute walk test.
  The test will be performed in an isolated room in order to avoid noise or external stimuli which can affect performance. The stepper will be placed near a door and the patient was allowed to put a hand on it if out of balance or exhausted. The height of the step will be fixed to 20 cm. A step was defined as the rise and lowering of one foot. The patient was informed of the time each minute. No other encouragement was given. Heart rate and transcutaneous oxygen saturation will be continuously recorded by a pulse oximetry.

SUMMARY:
Chronicle obstructive pulmonary disease is a worldwide cause of mortality and morbidity. This systemic disease progressively leads to dyspnea, muscle wasting and exercise capacity impairment.

Pulmonary rehabilitation is a cornerstone in the management of these systemic effects. Unfortunately, access to pulmonary rehabilitation is limited for many people who would benefit from it, primarily because of a lack of pulmonary rehabilitation and assessment centers. Optimal assessment should include cardiopulmonary exercise testing to determine both the optimal training settings as well as any cardiopulmonary contraindications to pulmonary rehabilitation. However, this is not available in most centers and when it is, consultations are limited. Therefore, pulmonary rehabilitation is often delayed for several weeks and patients can lose motivation.

In order to promote pulmonary rehabilitation, the incremental cardiopulmonary exercise testing could be replaced by field tests to individualize pulmonary rehabilitation prescription.

The 6-minute stepper test is a new field tool. Its sensitivity and reproducibility have previously been reported in patients with chronicle obstructive pulmonary disease. It is easy to set up in the clinical setting and could be used to individualize pulmonary rehabilitation.

The aim of this study was to develop and validate a prediction equation to set rehabilitation intensity for patients with severe to very severe chronicle obstructive pulmonary disease attending pulmonary rehabilitation, with the use of a simple, readily available field test. Therefore the investigators sought to determine, if it exists, a relationship between the plateau heart rate from the first and last 3 minutes of the 6-minute stepper test and the heart rate from the first ventilatory threshold from the cardiopulmonary exercise testing in order to individualize pulmonary rehabilitation in patients with severe to very severe chronicle obstructive pulmonary disease.

DETAILED DESCRIPTION:
Experimental design:

The validation of the six-minute stepper test to prescribe endurance training in severe to very severe chronicle obstructive pulmonary disease involves two steps :

1. Patients with severe to very severe chronicle obstructive pulmonary disease who performed an incremental cardiopulmonary exercise testing and are referred to pulmonary rehabilitation will be approached to participate in the study.

   Eligible patients who agree to participate in the study and sign informed consent will perform two six-minute stepper test. Their performance and heart rate (first and last 3minutes) will be compared with those obtained at the first ventilatory threshold from the previously performed incremental cardiopulmonary exercise testing (usually used for the prescription of endurance training in pulmonary rehabilitation) using multiple regression in order to derive a predictive equation.
2. The validity of this predictive equation will be assessed in an independent cross-validation group issued from a completed multicenter observational study (NCT03244137). This cross-validation group will be formed with those patients of this cohort who performed both the incremental cardiopulmonary exercise testing (and had a determined first ventilatory threshold) and the six-minute stepper test. The heart rate prescription for endurance training from the direct measurement of the the first ventilatory threshold will be compared to the heart rate derived from the 6minute-stepper test using the predictive equation determined in step 1. Data will be compared using the mean absolute difference between both prescriptions and a Bland-Altman analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans ;
* Chronicle obstructive pulmonary disease stage III/IV (FEV1 < 50%) ;
* Weight ≤ 90kg ;
* Eligible for pulmonary rehabilitation ;
* A first ventilatory threshold has been identified during a previously performed incremental cardiopulmonary exercise testing.

Exclusion Criteria:

* Pregnant woman or likely to be ;
* Patient under guardianship ;
* Contraindication to cardiopulmonary exercise testing ;
* Patient medically treated with heart rate modulator (excluding oral B2-agonist) ;
* Patient treated with pacemaker or defibrillator ;
* History of lower limb impairment (i.e. peripheral artery disease, orthopedic disorder etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe to very severe chronicle obstructive pulmonary disease reffered for pulmonary rehabilitation.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Relation between plateau heart rate (bpm) from the first and last 3 minutes of the 6-minute stepper test and heart rate (bpm) from first ventilatory threshold from cardiopulmonary exercise testing. | Heart rate (bpm) will be assessed during cardiopulmonary exercise testing with electrocardiogram. During the 2 6-minute stepper test, heart will be assessed with oximeter. All theses tests wil be carried out in a total time frame of 3 month maximum.
  Outcome (heart rate) during different tests will be continuously recorded. Relation will be adjusted for age and step count.

SECONDARY OUTCOMES:
Relation between minimal SpO2 (%)from the 6-minute stepper test and SpO2 (%) from first ventilatory threshold from cardiopulmonary exercise testing. | SpO2 will be assessed with oximeter. All theses tests wil be carried out in a total time frame of 3 month maximum.
  Outcome (SpO2 (%)) during different tests will be continuously recorded. Relation will be adjusted for age en step count.
Diastolic blood pressure (mmHg) before and after every 6-minute stepper test using electrical blood pressure device. | The outcome will be assessed before and after every 6-minute stepper test. The 2 6-minute stepper test will be carried out the same day (minimum 20 minute of rest between each test) for a total time frame of 1 day.
Systolic blood pressure (mmHg) before and after every 6-minute stepper test using electrical blood pressure device. | The outcome will be assessed before and after every 6-minute stepper test. The 2 6-minute stepper test will be carried out the same day (minimum 20 minute of rest between each test) for a total time frame of 1 day.
Steps during 6-minute stepper test using stepper device. | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
Dyspnea using the Borg scale. | Dyspnea will be assessed at the end of every tests for a total time frame of 2 hours.
  Borg scale range from 0 (no breathlessness) to 10 (maximal breathlessness)
Lower limb fatigue using the Borg scale. | Lower limb fatigue will be assessed at the end of every tests for a total time frame of 2 hours.
  Borg scale range from 0 (no breathlessness) to 10 (maximal breathlessness)

CONTACTS AND LOCATIONS:
Overall Officials: David Debeaumont, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Catherine Tardif, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Antoine Cuvelier, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.; Tristan Bonnevie, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Catherine Viacroze, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Bouchra Lamia, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Jean Quieffin, MD, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Guillaume Prieur, PT, MsC, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Clément Médrinal, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France; Pierre-Alexandre Hauss, MD, Study Chair — Service de pneumologie, Centre Hosptalier Intercommunal Elbeuf-Louviers-Val de Reuil
Locations (4):
- France (4):
  - ADIR Association, Bois-Guillaume
  - Centre Hostalier Intercommunal Elbeuf-Louviers-Val de Reuil, Elbeuf
  - Groupe Hospitalier du Havre, Le Havre
  - Centre Hospitalier de Morlaix, Morlaix

IPD SHARING:
Plan to Share IPD: No